CLINICAL TRIAL: NCT00063219
Title: A Phase 2, Open-label Study of MAC-321 Administered Intravenously as a Single Agent for the Treatment of Non-small Cell Lung Cancer Refractory to Platinum-based Therapy
Brief Title: Study Evaluating MAC-321 in Non-small Cell Lung Cancer Refractory to Platinum-based Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 3128K1-201
Record Dates: First submitted 2003-06-23; First posted 2003-06-25 (Estimated); Last update posted 2009-08-21 (Estimated); Status verified 2009-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Lung Neoplasms
Keywords: Non-Small-Cell Lung Carcinoma; Lung Cancer; Cancer of Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — MAC321

INTERVENTIONS:
Drug: MAC-321

SUMMARY:
This non-randomized, open-label clinical trial is designed to determine safety and clinical activity of a new chemotherapeutic agent, MAC-321, when given intravenously to patients with non-small cell lung cancer. Clinical activity will be evaluated by determining the percentage of patients with an objective tumor response after treatment with MAC-321. Patients must have been previously treated with a platinum-containing chemotherapy regimen.

A total of 96 patients will be enrolled in this trial. Eligible patients will receive MAC-321 intravenously every 3 weeks for up to a total of 6 courses of treatment. All patients will receive MAC-321 at the same dose. MAC-321 is an experimental drug, and is not offered outside of this research trial.

ELIGIBILITY:
Inclusion Criteria:

* Recurrence of non-small cell lung cancer after at least 1 prior chemotherapy regimen containing a platinum agent
* Recovery from all acute side effects of prior therapies (with the exception of hair loss)
* Adequate bone marrow, liver, and kidney function

Exclusion Criteria:

* More than 2 prior chemotherapy regimens for treatment of advanced or metastatic non-small cell lung cancer. (Treatment given in conjunction with surgery will not be included in the maximum of 2 prior regimens)
* Radiation therapy, chemotherapy or any other anticancer therapy within 28 days of beginning study
* Symptomatic brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (13):
- United States (13):
  - Los Angeles, California
  - Lexington, Kentucky
  - Baltimore, Maryland
  - Worcester, Massachusetts
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - New York, New York
  - Charlotte, North Carolina
  - Cleveland, Ohio
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Nashville, Tennessee